CLINICAL TRIAL: NCT01548937
Title: Serotonin Transporter Density in Late-life Depression With and Without Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 98-2132A
Record Dates: First submitted 2011-12-29; First posted 2012-03-08 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Melancholia
Keywords: I-123 ADAM Serotonin transporter imaging
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I-123 ADAM (Experimental): I-123 ADAM Serotonin transporter imaging
  Interventions: Drug: I-123 ADAM

INTERVENTIONS:
Drug: I-123 ADAM — This study will recruit a total of 40 evaluable subjects (20 cognitively depressive, and 20 AD depressive), Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping.
  Safety measurement will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.

SUMMARY:
This study will recruit a total of 40 evaluable subjects (20 cognitively depressive, and 20 AD depressive); each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping.

Safety measurement will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.

This study is expected to be completed in a period of 3 years.

DETAILED DESCRIPTION:
Depression and dementia are the two common psychiatric disorders in the elder subjects. Alzheimer's disease (AD) is the most frequent cause of dementia and about 20% of them have depression. Depression subjects are associated with more rapid cognitive decline, a poorer response to treatment. Post mortem study showed close relationship between AD and disruptions of the serotonergic system, including loss of serotnergic neurons at brain stem. However, the alternations in presynaptic serotonin function relative to demented or non-demented subjects remain to be investigated in living subjects. In this study, the investigators will collect 40 elder subjects (i.e., age above or equal to 50 years old). The serotonin transporter activity will be compared between subjects with or without dementia using I-123 ADAM images. The single photon emission tomography (SPECT) will be compared to recent (within 6 months) F-18 FDG PET images for further investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients may be enrolled in the AD depressive group if they:

   * Are males or females at least 50 years of age;
   * Fulfilled the DSM-IV criteria for Major depressive disorder (APA, 1994) by MINI interview.
   * Meet the NINCDS/ADRDA(National institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association) criteria for probable AD
   * A Mini Mental State Examination (MMSE) score at screening between 10 and 24 inclusive;
   * Give informed consent. If the patient is incapable of giving informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
2. Patients may be enrolled in the cognitively depressive group if they:

   * Are males or females at least 50 years of age;
   * Fulfilled the DSM-IV criteria for Major depressive disorder (APA, 1994) by MINI interview.
   * Memory function above the lower normal limits (i.e. 1.5 SD above the mean) on tests for episodic memory.
   * Clinical Dementia Rating = 0. Memory Box score must be 0.
   * Cognitively normal, based on an absence of significant impairment in cognitive functions or ADL.
   * A MMSE score at screening > 24 for those with education level of 6 years or above and > 17 for those are illiterate;
   * Give informed consent.

Exclusion Criteria:

* Pregnant or becoming pregnant during the study (as documented by pregnancy testing at screening or at any date during the study according to the PI discretion) or current breast feeding.
* Conditions affecting brain structure or function (e.g., stroke, diabetes, head trauma, depression) or use of cognitively
* Substance abuse.
* Alcohol dependence

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the differences of serotonin transporter activity among depressive patient with or without dementia. | three years
  To expand the database of I-123 ADAM SPECT imaging in AD depressive and cognitively depressive patients to refine the definition of a positive scan in patient with AD and MDD.

SECONDARY OUTCOMES:
Evaluate the relationship between the serotonin transporter activity and F-18 FDG PET image patter. | three years
  To expand the safety database of I-123 ADAM SPECT imaging Safety variables include adverse event count, lab parameters, vital signs, and ECG. Comparison will be generally made to baseline, as appropriate.